CLINICAL TRIAL: NCT00767221
Title: Oral Treatment With PL-56 in Patients With IgA Nephropathy - an Explorative Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Calliditas Therapeutics AB (Industry)
Collaborators: Archimedes Development Ltd (Industry)
Responsible Party: Johan Häggblad, Pharmalink AB
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U-03-003
Record Dates: First submitted 2008-10-05; First posted 2008-10-07 (Estimated); Last update posted 2009-04-21 (Estimated); Status verified 2009-04

CONDITIONS: IGA Nephropathy
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Budesonide; Anti-Inflammatory Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): The patient is his own control. Endpoint variables are measured before, during and after treatment.
  Interventions: Drug: Budesonide

INTERVENTIONS:
Drug: Budesonide — 8 mg PL-56 once daily for six months
  Other Names: Nefecon, PL-56 (topical acting, anti-inflammatory agent)

SUMMARY:
The study will investigate the effect of PL-56 on albumin leakage and renal function (glomerular filtration rate) in patients with IgA nephropathy. It will also assess the safety of treatment with PL-56.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Female or male patient > 18 years
* Biopsy-verified IgA nephropathy
* Proteinuria: U-albumin >500 mg/24 h
* S-creatinine < 200 umol/L
* A minimum of four available sample results (U-albumin and S-creatinine) prior to inclusion in the study.

Exclusion Criteria:

* Severe gastrointestinal disorders which may impair drug effect, or other conditions which could modify the effect of the trial drug as judged by the investigator
* Consumption of an investigational drug within 30 days prior to enrolment
* Unacceptable blood pressure (treated or untreated), defined as a systolic value >150 mm Hg and/or diastolic >90 mm Hg
* Hyperlipidaemia defined as unacceptable levels of lipids according to the discretion of the Investigator
* Patients in whom an ACE inhibitor was introduced/changed during the last three months prior to enrolment
* Patients treated with immuno-suppressive drugs
* Patients unable to take oral medication
* Severe liver disease (defined as ASAT and/or ALAT and/or gamma-GT above twice the normal value).
* Uncontrolled (treated or untreated) congestive heart failure as judged by the Investigator
* Patients with diabetes
* Patients with current malignancy or history of malignancy during the last three years
* History or presence of psychological or psychiatric illness which may interfere with the patient´s ability to adhere to the protocol
* Alcohol or drug abuse (present)
* Patients unwilling to meet the requirements of the protocol
* Other medical or social reasons for exclusion at the discretion of the Investigator
* Use of drugs inhibiting the cytochrome P-450 enzyme CYP3A4 (including grape fruit juice)
* Kidney transplanted patients
* For women only: pregnant or breast feeding; unwilling to use adequate contraception during the study (only women of childbearing potential)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2005-10; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
U-albumin | 6(treatment)+3(follow-up) months

SECONDARY OUTCOMES:
GFR and safety | 6(treatment) + 3(follow-up) months

CONTACTS AND LOCATIONS:
Overall Officials: Bengt Fellström, MD, PhD, Principal Investigator — Uppsala University Hospital, Dept. of Medicine
Locations (3):
- Sweden (3):
  - Linköping University Hospital, Linköping
  - Huddinge University Hospital, Stockholm
  - Uppsala University Hospital, Uppsala